CLINICAL TRIAL: NCT05461729
Title: TIMELY Prospective Study
Acronym: TIMELY
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dr. Boris Schmitz (Other)
Collaborators: European Commission (Other); University of Amsterdam (Other); Technische Universität Dresden (Other); MEDIZINISCHE UNIVERSITAT GRAZ (Unknown); Stichting Katholieke Universiteit (Other); Foundation for Research and Technology - Hellas (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Boris Schmitz, Primary Researcher Department of Rehabilitation Sciences, University of Witten/Herdecke
Organization: University of Witten/Herdecke (Other)
Other Study IDs: TIMELY_P01
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease
Keywords: Cardiac Rehabilitation; Telemedicine; Healthy Lifestyle; Preventive Programs; Artificial Intelligence; Predictive Medicine; Continuum of Care; Maintenance; Aftercare; eHealth; mHealth
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease: Patients with Coronary Artery Disease

SUMMARY:
Brief Summary:

Cardiac rehabilitation (CR) is a multi-factorial intervention, designed to limit the physiological and psychological effects of cardiovascular disease such as coronary artery disease (CAD), manage symptoms, and reduce the risk of future cardiovascular events. CR is a structured program not only addressing CAD but also comorbidities including hypertension, dyslipidemia, diabetes and obesity as well as other risk factors. CR aims at long-term lifestyle changes to reduce modifiable risk factors, and it's success depends on a large number of interacting variables including biological, psychological and social factors. Recently, the importance of patient-centered approaches to secondary prevention and CR success has been underlined but intra-individual factors and their interactions are not well understood. The TIMELY prospective study aims to collect high-resolution data for data mining and artificial intelligence machine learning models to identify dependencies between factors and predict favorable outcomes of CR. Data collection will include data documented during controlled center-based CR as well as remote-measurement of physical activity data, (central) blood pressure and pulse wave analysis as well as long-term ECG data during a 6-months period after discharge. Follow-up assessments will be performed at least at 6 months and at 12 months after discharge.

Main objectives of the study:

1. To examine uptake and adherence to a healthy lifestyle (i. e. adherence to CR guidelines in CAD) and the effects on long-term outcomes.
2. To identify potentially mediating mechanisms and predictive factors for long-term CR success in CAD.
3. To investigate acceptance of different eHealth components as well as expectations and needs among CAD patents in CR.

ELIGIBILITY:
Inclusion Criteria:

Coronary Artery Disease (CAD) patients after myocardial infarction (STEMI/NSTEMI) and/or angioplasty and/or Percutaneous Coronary Intervention (PCI) and/or coronary artery bypass graft surgery who participate in phase II Cardiac Rehabilitation (CR).

Exclusion Criteria:

* Incapability to give informed consent
* Conditions that prevent patients from participation in CR including unstable coronary or cerebrovascular conditions and acute infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary Artery Disease (CAD) patients participating in phase II Cardiac Rehabilitation (CR).
Sampling Method: Non-Probability Sample
Enrollment: 612 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiorespiratory Fitness (CRF) | Baseline, week 3, and week 24
  CRF will be measured as maximal oxygen uptake (VO2max) determined by spiroergometry
Change in risk of mortality | Baseline, week 3, and week 24
  Risk of mortality will be determined using the validated biomarker risk score COROPREDICT
Number of patients with major adverse cardiac and cerebrovascular events (MACCE) | Baseline to week 48
  Number of patients with death, myocardial infarction, stent thrombosis, stroke or transient ischemic attack, urgent revascularization, and major bleeding

SECONDARY OUTCOMES:
Physical activity (PA) | Baseline, week 3, week 24, and week 48
  PA will be measured by validated BSA questionnaire (Bewegungs- und Sportaktivität) and expressed as metabolic equivalents
Daily step count | Baseline to week 24
  Steps will be measured using electronic devices such as wrist-worn activity trackers
Weekly number and duration of physical activities | Baseline to week 24
  Number and duration of physical activities will be measured using electronic devices such as wrist-worn activity trackers
Resting heart rate | Baseline to week 24
  Resting heart rate will be measured using electronic devices such as wrist-worn activity trackers
Sleep duration | Baseline to week 24
  Sleep duration will be measured using electronic devices such as wrist-worn activity trackers
Physiological stress | Baseline to week 24
  Physiological stress will be measured using electronic devices such as wrist-worn activity trackers
Blood pressure | Baseline to week 24
  Central and peripheral systolic and diastolic blood pressure will be measured using automatic upper-arm sphygmomanometers. Data transmitted by telemetry.
Arterial pressure wave propagation/reflection characteristics | Baseline to week 24
  Arterial pressure wave propagation/reflection characteristics will be measured using automatic upper-arm tonometry. Data transmitted by telemetry.
Cardiac arrhythmia | Baseline to week 24
  Cardiac arrhythmia will be measured using three-channel Holter ECG.
Body composition | Baseline, week 3, and week 24
  Body composition including fat mass, muscle mass, and visceral fat area will be measured by bioimpedance analysis.
Muscle strength | Baseline, week 3, and week 24
  Arm and leg extension and flexion strength will be measured using Isokinetic devices
Muscle function | Baseline, week 3, and week 24
  Muscle function will be measured by 30-second chair rise test
Submaximal exercise capacity | Baseline, week 3, and week 24
  Submaximal exercise capacity will be measured using 6-min walking test
Habit formation | Baseline, week 3, week 24, and week 48
  Habit formation will be assessed using validated questionnaire for the "Self-Report Behavioural Automaticity Index (SRBAI)".
Nicotine dependence | Baseline, week 3, week 24, and week 48
  Nicotine dependence will be assessed using the Fagerström questionnaire
Cardiac Self-Efficacy | Baseline, week 3, week 24, and week 48
  Cardiac Self-Efficacy will be assessed using the validated "Cardiac Self-Efficacy Scale (CSE)"
Impact of disease | Baseline, week 3, week 24, and week 48
  Impact of disease will be assessed using the "brief illness perception (IPQ-9)" questionnaire .
General wellbeing | Baseline, week 3, week 24, and week 48
  General wellbeing will be assessed using the "Positive And Negative Affect Scale (PANAS)" questionnaire .
Fear of Activity/ Kinesiophobia | Baseline, week 3, week 24, and week 48
  Fear of Activity/ Kinesiophobia will be assessed using the modified "Fear of Activity Scale (FActS)".
Depression | Baseline, week 3, week 24, and week 48
  Depression will be assessed using the modified "Patient Health Questionnaire (PHQ-9)".
General anxiety | Baseline, week 3, week 24, and week 48
  General anxiety will be assessed using the "7-item General Anxiety Scale (GAD-7)".
Health-related quality of life | Baseline, week 3, week 24, and week 48
  Health-related quality of life will be assessed using the "RAND 36-Item Health Survey (SF-36)".
General quality of life | Baseline, week 3, week 24, and week 48
  Quality of life will be assessed using the "5-level EQ-5D (EQ-5D-5L) health status measure".
Wellbeing | Baseline, week 3, week 24, and week 48
  Wellbeing will be assessed using the "WHO-5 Well-Being Index".
Perceived stress | Baseline, week 3, week 24, and week 48
  Perceived stress will be assessed using the "Perceived Stress Scale (PSS-4)".
Optimism/ Pessimism | Baseline, week 3, week 24, and week 48
  Optimism/ Pessimism will be assessed using the modified "Life Orientation Test (LOT-R)".
Conscientiousness | Baseline, week 3, week 24, and week 48
  Conscientiousness will be assessed using the "The Big Five Inventor (BFI-10)".
Psychological flexibility | Baseline, week 3, week 24, and week 48
  Psychological flexibility will be assessed using the psychometric properties of the "Acceptance and Action Questionnaire-I (AAQ-II)".
Negative Affectivity | Baseline, week 3, week 24, and week 48
  Standard assessment of negative affectivity, social inhibition, and Type D personality (DS-14)
Trait anger | Baseline, week 3, week 24, and week 48
  Trait anger will be assessed using the "State-Trait Anger Expression Inventory-2 ("TAI-10/STAXI-2").
Religiousness/ spirituality | Baseline, week 3, week 24, and week 48
  Religiousness/ spirituality will be assessed using the "Spiritual and Religious Attitudes in Dealing with Illness (GrAw-7/ SpREUK-15)" questionnaire.
Fatigue | Baseline, week 3, week 24, and week 48
  Fatigue will be assessed using the "The Multidimensional Fatigue Inventory (MFI20)".
Psychological situation in the working environment | Baseline, week 3, week 24, and week 48
  Psychological situation in the working environment will be assessed using the "The effort-reward imbalance model (ERI10+6)".
Work requirements and workload | Baseline, week 3, week 24, and week 48
  Work requirements and workload will be assessed using the "Workability Index (WAI)".
Social support | Baseline, week 3, week 24, and week 48
  Social support will be assessed using the short "Perceived Social Support Questionnaire (F-SozU K6)".
Relationship satisfaction | Baseline, week 3, week 24, and week 48
  Relationship satisfaction will be assessed using the "Quality of Marriage Index (QMI)".

OTHER OUTCOMES:
Needs and requirements for eHealth in cardiac rehabilitation | Week 3
  Needs and requirements for eHealth in cardiac rehabilitation will be assessed using questionnaires, interviews, and focus groups.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Schmitz, PhD, Principal Investigator — University of Witten/Herdecke, Dpt. Rehabilitation Sciences
Locations (1):
- Klinik Königsfeld, Ennepetal, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmitz B, Wirtz S, Sestayo-Fernandez M, Schafer H, Douma ER, Alonso Vazquez M, Gonzalez-Salvado V, Habibovic M, Gatsios D, Kop WJ, Pena-Gil C, Mooren F. Living Lab Data of Patient Needs and Expectations for eHealth-Based Cardiac Rehabilitation in Germany and Spain From the TIMELY Study: Cross-Sectional Analysis. J Med Internet Res. 2024 Feb 22;26:e53991. doi: 10.2196/53991. PMID 38386376